CLINICAL TRIAL: NCT03341000
Title: Pilot Study to Examine the Feasibility of the DISCSS™
Brief Title: Pilot Study to Examine the Feasibility of the Dynamic Interferential Spinal Cord Stimulation System™ (DISCSS™)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Meagan Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: DISCSS 01
Record Dates: First submitted 2017-10-27; First posted 2017-11-14 (Actual); Results first posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Intervention Model Description: prospective, multi-center, open-label, feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- DISCSS Device (Experimental): This pilot feasibility study will explore and help determine optimal settings and configuration of the DISCSS™ System with patients that have completed a percutaneous trial with a commercially available SCS trial system within the first 3-5 days of the current study.
  Interventions: Device: DISCSS Device

INTERVENTIONS:
Device: DISCSS Device — This pilot feasibility study will explore and help determine optimal settings and configuration of the DISCSS™ System with patients that have completed a percutaneous trial with a commercially available SCS trial system within the first 3-5 days of the current study.

SUMMARY:
This study evaluates use of DISCSS vis SCS. Thirty (30) patients with back pain greater than leg pain who were candidates for Spinal Cord Stimulation (SCS) and have successfully completed a percutaneous trial with a commercially available SCS system will be trialed with a 3-4 day exposure to the investigational DISCSS™ device. The trial will be conducted at 3-5 U.S. centers. The percutaneous trial leads from the commercial system will be connected to the External Pulse Generator of the DISCSS™ Trial System and the patients will be trialed for an additional three-four days.

DETAILED DESCRIPTION:
This investigation will be performed as a prospective, multicenter, open-label feasibility study. Thirty (30) patients with back pain greater than leg pain who were candidates for Spinal Cord Stimulation (SCS) and have successfully completed a percutaneous trial with a commercially available SCS system will be trialed with a 3-4 day exposure to the investigational DISCSS™ device. The trial will be conducted at 3-5 U.S. centers. The percutaneous trial leads from the commercial system will be connected to the External Pulse Generator of the DISCSS™ Trial System and the patients will be trialed for an additional three to four days. The investigational product for this feasibility trial will be the DISCSS™ system, not the commercially available trial SCS system. Exposure to the commercially available trial SCS system will be considered background therapy. The purpose of the background therapy phase is to establish baseline pain levels and determine patients' eligibility to continue to the investigational phase of the trial using the DISCSS™ SCS phase of the trial. Pain assessment and complications data from the commercial spinal stimulation system will be collected during the background therapy phase. The pain and complications data from the background therapy phase will not be analyzed in terms of the study endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 21 years and less than 80 years
2. Has a diagnosis of chronic neuropathic pain of trunk and limbs
3. Is eligible for and participating in a spinal cord stimulation trial of a commercially available SCS trial system. Subjects will be evaluated at the end of the background Commercial SCS Device phase for complications and appropriateness to continue to the investigational phase with the DISCSS™ system. Complications from the background phase with the commercial SCS device may include, but are not limited to unusual pain or discomfort during the trial stimulation, local skin reactions or infection at the implant site.
4. Has a Back Pain Score of minimum intensity 5.0 on a Numeric Rating Scale (NRS)
5. Has an NRS Back Pain Score that is greater than both Leg Pain Scores
6. Is not a candidate for revision surgery
7. Has completed a minimum of 6 weeks of conservative therapy (physical therapy, anti-inflammatory medications, or similar therapies) with limited or no reduction in back pain
8. Is willing to adhere to the warnings associated with the DISCSS™ system
9. Is willing to halt and/or modify the use of all prescription and over-the-counter analgesics per the Investigator's direction during study participation
10. Is capable of providing written informed consent
11. Is able to comply with the requirements of study visits, follow-up phone visits and self-assessment questionnaires

Exclusion Criteria:

1. Is a poor surgical candidate by determination of the Investigator
2. Is unable to operate or understand the use of the commercial or investigational Spinal Cord Stimulator systems
3. Has an active systemic infection
4. Has exposure to shortwave, microwave or ultrasound diathermy at home or at work
5. Has occupational exposure to high levels of non-ionizing radiation such as radio or cell phone transmission stations, facilities using radiofrequency heat sealers or induction heaters, or electric power infrastructure controlled environments
6. Has an implanted cardiac system (e.g. pacemakers)
7. Is currently participating in another clinical study
8. Is currently pregnant or lactating, or not using adequate birth control
9. Has any untreated major psychiatric comorbidity
10. Has serious drug-related behavioral issues per Investigator's assessment
11. Has a bleeding complication or coagulopathy
12. Requires concurrent use of anticoagulant therapy such as heparin, warfarin, rivaroxaban, dabigatran, apixaban, edoxaban, enoxaparin, fondaparinux
13. Is immunocompromised and at risk for infection
14. Has insulin-dependent diabetes not controlled through diet and/or medication
15. Has chronic pain related to malignancy
16. Is otherwise determined, based on the opinion of the Investigator to be an unsuitable candidate for this study

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Pain Treatment Centers, Ocala, Florida
  - Sarasota Memorial Pain Care Center, Sarasota, Florida
  - The Brigham and Women's Hospital, Boston, Massachusetts
  - Neuromodulation Specialists, LLC, Pascagoula, Mississippi
  - Precision Spine Care, Tyler, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- DISCSS Device: This pilot feasibility study will explore and help determine optimal settings and configuration of the DISCSS™ System with patients that have completed a percutaneous trial with a commercially available SCS trial system within the first 3-5 days of this study.
  DISCSS Device: This pilot feasibility study will explore and help determine optimal settings and configuration of the DISCSS™ System with patients that have completed a percutaneous trial with a commercially available SCS trial system within the first 3-5 days of this study.
Period: Overall Study
Arm/Group | DISCSS Device
Started | 18
Completed | 17
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- DISCSS Device: This pilot feasibility study will explore and help determine optimal settings and configuration of the DISCSS™ System with patients that have completed a percutaneous trial with a commercially available SCS trial system.
  DISCSS Device: This pilot feasibility study will explore and help determine optimal settings and configuration of the DISCSS™ System with patients that have completed a percutaneous trial with a commercially available SCS trial system.
Arm/Group | DISCSS Device
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
Height [Mean (Standard Deviation); unit: Inches] | 67.6 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Day 1) to Visit 5 in Back Pain.
Description: Change from baseline (day 1) to visit 5 (day 10-11) in patient-reported pain intensity, measured on a Numeric Rating Scale (NRS) ranging from 0 (no pain) to 10 (worst pain).
Time Frame: Baseline to visit 5
Population: Intent to treat.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DISCSS Device
Number analyzed (Participants) | 17
score on a scale
  Overall | -4.2 (2.3)
  Lower Extremity | -3.9 (2.5)
  Back | -4.4 (2.3)

2. Secondary Outcome: Incidence of Adverse Events
Description: Incidence of adverse events arising from the DISCSS treatment phase
Time Frame: Visit 4 (Day 6-7), and Visit 5 (Day 10-11)
Population: All enrolled subjects.
Measure: Number; unit: Adverse Events
Arm/Group | DISCSS Device
Number analyzed (Participants) | 18
Adverse Events
  Serious Adverse Event | 1
  Adverse Event | 6

3. Secondary Outcome: Patient Satisfaction
Description: Patient-reported device efficacy and device stimulation sensation as captured on a study-specific, subject satisfaction Questionnaire.
Time Frame: Visit 5 (Day 10-11)
Population: Intent to treat.
Measure: Count of Participants; unit: Participants
Arm/Group | DISCSS Device
Number analyzed (Participants) | 17
Participants
  Very Satisfied | 9
  Satisfied | 4
  Somewhat Satisfied | 3
  Dissatisfied | 1

ADVERSE EVENTS:
Time Frame: Visit 1 (Day 1), Visit 2 (Day 0-3) and 3 (Day 4 - 5), Visit 4 (Day 6-7), and Visit 5 (Day 10-11)
Groups:
- DISCSS Device: 3-5 days of DISCSS following the completion of a 3-5 day trial with a commercially available SCS system.
- SCS System: 3-5 day trial with a commercially available SCS system
Arm/Group | DISCSS Device | SCS System
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/18
Other Adverse Events (participants affected / at risk) | 5/18 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DISCSS Device (N=18) | SCS System (N=18)
Percutaneous Trial Lead Fracture (Product Issues) | 1 (1) | 0 (0) — Fracture of commercial trial lead upon removal at the end of the DISCSS trial (visit 5).
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DISCSS Device (N=18) | SCS System (N=18)
Increased Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Burning/Shocking (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lead Migration (Product Issues) | 2 (2) | 0 (0)
Painful Stimulation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT03341000/Prot_000.pdf